CLINICAL TRIAL: NCT06766955
Title: Prevalence of Lower Cross Syndrome Among Female College Students and Its Relation With Dysmenorrhea
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Farida Bakr Mohamed, Principal investigator, Cairo University
Other Study IDs: P.T.REC/012/005378
Record Dates: First submitted 2025-01-04; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Cross Syndrome
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- female college students: 140 Medical and Non-Medical Female students participated in this study. They were selected randomly from Cairo University and the British university in Egypt.

INTERVENTIONS:
Other:

SUMMARY:
The purpose of the study is to find out the prevalence of lower cross syndrome among female college students and its relation with dysmenorrhea.

DETAILED DESCRIPTION:
In individuals with lower cross syndrome (LCS), there is often a notable tightness in the hip flexors and the lower back musculature, which is typically accompanied by a corresponding weakness in the abdominal muscles and the gluteus maximus. This imbalance is not merely a matter of discomfort; it fundamentally disrupts the normal distribution of biomechanical forces within the lower back. When the muscles that support the pelvis and spine are not functioning optimally, it can lead to altered movement patterns and increased strain on the lumbar region.

The positioning of the uterus can also be adversely affected by this muscular imbalance. Anterior or posterior displacement of the uterus can occur as a result of the altered pelvic alignment associated with LCS. This displacement can create additional tension within the surrounding soft tissues and muscles, leading to a cascade of physiological responses.

One notable consequence of this tension is the excessive secretion of prostaglandins, which are hormone-like substances that play a key role in the regulation of inflammation and pain. Elevated levels of prostaglandins are often linked to dysmenorrhea, or painful menstruation, which can further exacerbate discomfort and impact the daily lives of those affected.

To date, there is only one previous study in India investigating the prevalence of LCS among female college students and its relation with dysmenorrhea. There is lack of literature evidence, which can show the prevalence of LCS among female college students in Egypt. So, this study aims to fill a critical gap in existing literature by providing valuable insights into the prevalence and associated factors of LCS in this population in Egypt.

ELIGIBILITY:
Inclusion Criteria:

* They were virgin, healthy female college students.
* They had regular menstruation (3-8 days in duration, with 21-35 days in-between).
* Their ages ranged from 18 to 25 years old.
* Their body mass index (BMI) will range from 18 to 24.9 Kg/m2.
* Their waist- hip ratio was less than (0.8).

Exclusion Criteria:

* History of back or lower limb surgery
* Trauma to back or lower extremity
* Rheumatoid arthritis
* Spinal deformity such as kyphosis and scoliosis.
* Any neurological disease
* Uncooperative volunteers.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Medical and Non-Medical Female students participated in this study. They were selected randomly from Cairo University and private universities in Cairo.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2025-02-25 (Estimated); Study Completion 2025-03-13 (Estimated)

PRIMARY OUTCOMES:
Measurement of iliopsoas muscle length | 6 weeks
  The Thomas test is used to assess the hip flexion Tightness. Position: The measurement of iliopsoas muscle length involved the subject lying supine on a plinth with one thigh protruding while the examiner checks for excessive lordosis. The non-tested hip is flexed and held close to the chest to stabilize the pelvis and flatten the lumbar spine. Using a universal goniometer, the examiner measures the iliopsoas length on the opposite side. The fulcrum is placed above the greater trochanter, the movable arm parallel to the femoral shaft, and the stationary arm parallel to the plinth. If the hip flexion angle exceeds 15 degrees, the patient's straight leg rises off the table and a muscle stretch end feel will be felt, the iliopsoas is considered tight.
Measurement of length of spinal extensors muscle | 6 weeks
  The length of the spinal extensor muscles will be measured by modified Schober test while a female college student standing and her back facing the examiner. A reference line is marked at the intersection of the Venus dimples (Posterior superior iliac spine PSIS) on her lower back, with additional lines drawn 10 cm above and 5 cm below this point. The student then bends forward, and the examiner measured the increase in distance between these points using a measuring tape. The outcome measure is calculated by determining the differences between these points
Measurement of strength of abdominal muscle | 6 weeks
  In this procedure, females are placed in a supine position with different arm placements based on the grade. The examiner stands beside the table at the chest level to ensure the scapula clears the table. The patient is asked to assume the end position by flexing their trunks fully, curling up until the scapula is off the table. They were guided with the instruction, "Tuck your chin and lift your head, shoulders, and arms off the table, as if doing a sit-up and hold it." (Magee, 2002).
  The gradings of this test are:
  Normal 5= Hands behind neck, until scapulae clear table 20-30sec hold. Good 4= Arms crossed over chest, until scapulae clear table 15-20sec hold. Fair 3= Arms straight, until scapulae clear table 10-15 sec held. Poor 2= Arms extended, towards knees, until top of scapulae lift from table 1-10 sec hold.
  Trace 1= Unable to raise more than head off table.
Measurement of gluteus Maximus strength | 6 weeks
  The subject is placed in prone with the hips straight and the knee flexed to 90 degrees. The student is asked to extend the hip, keeping the knee flexed. Anterior force is applied to the posterior thigh. The pelvis is stabilized during the movement. Both legs are tested.
  The grading of this test are:
  Normal 5 = indicates that the individual achieves complete hip extension and can maintain the end position against maximal resistance.
  Good 4 = signifies that hip extension is achievable and can be sustained against heavy to moderate resistance.
  Fair 3 = denotes the ability to complete full hip extension and maintain the end position, although no resistance is applied.
  Poor 2 = reflects the capacity to perform the full range of hip extension while in a side-lying position.
  Trace 1 = is characterized by palpable contractions of the gluteus maximus, which manifest as a narrowing of the gluteal crease, without any observable movement at the joint.

SECONDARY OUTCOMES:
Assessment of menstrual symptoms | 6 weeks
  The Menstrual Distress Questionnaire (MEDI-Q) includes 25 items that cover symptoms related to menstruation, such as pain, discomfort, psychological or cognitive changes, and gastrointestinal issues. It evaluates the impact of these symptoms on daily functioning and quality of life during the menstrual phase and compares their frequency to the intermenstrual and premenstrual phases. The MEDI-Q provides scores for specific symptoms and four overall indices for a comprehensive assessment of menstrual distress. The MEDI-Q is a valid and reliable tool for assessing menstrual distress and its impact on psychological well-being. The items include subtitles ranging from 0 to 3. The total score ranges from 0 to 125. Lower score indicates lower menstrual symptoms and vice versa.

CONTACTS AND LOCATIONS:
Overall Officials: Amir A Gabr, Professor, Study Director — Cairo University; Dalia M. Kamel, Professor, Study Chair — Cairo University
Locations (1):
- Farida Bakr Mohamed, Cairo, Egypt